CLINICAL TRIAL: NCT06038747
Title: Investigating the Impact of Regular Self-monitoring and Reflecting on Affective Reactions Toward the Psychotherapist on Treatment Outcomes: A Randomized Controlled Trial Protocol.
Brief Title: Self-monitoring and Reflection's Impact on Psychotherapy Outcomes: A Trial Protocol.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Pavia (Other); European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-1067
Record Dates: First submitted 2023-09-06; First posted 2023-09-15 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Psychotherapy; Therapeutic Alliance; Psychological
Keywords: Therapeutic Relationship; Routine Outcome Monitoring; Self-Monitoring and Reflection; Psychotherapy Outcome; Client Feedback
MeSH Terms: interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial design. Allocation ratio of 1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual Psychotherapy + Self-Monitoring (Experimental): Participants in the intervention group will continue their regular individual psychotherapy sessions. Additionally, after each session, they will complete a brief postsession battery consisting of two scales on the affective reactions of the participants towards their therapist during session and read general feedback encouraging them to discuss their feelings and reflections with their therapist. This questionnaire aims to prompt reflection on the own experience of the therapeutic relationship.
  Interventions: Other: Self-Monitoring; Other: Individual Psychotherapy
- Individual Psychotherapy (Active Comparator): Participants in the control group will receive only treatment as usual (i.e., individual psychotherapy) sand and will not complete post-session questionnaires. Additionally, they will not receive any feedback at all encouraging them to discuss their emotional responses with their therapist during the session.
  Interventions: Other: Individual Psychotherapy

INTERVENTIONS:
Other: Self-Monitoring — The post-session battery consists of two self-report scales measuring both positive and negative affective reactions of the participants toward their therapist during the therapy session. The general feedback is a brief text that encourages participants to share and discuss their feelings and reflections with their therapist.
  Arms: Individual Psychotherapy + Self-Monitoring
Other: Individual Psychotherapy — Individual psychotherapy sessions

SUMMARY:
The primary objective of this randomized controlled trial is to examine the influence of a brief post-session battery, designed to foster patient self-monitoring and reflection on their emotional reactions toward their psychotherapist, on the quality of the therapeutic relationship and treatment outcomes.

DETAILED DESCRIPTION:
The quality of the therapeutic relationship is critical in determining psychotherapy outcomes. However, facilitating patients' self-awareness and reflection on their affective responses to their therapist remains understudied as a potential tool for enhancing this relationship and subsequent treatment outcomes. The primary objective of this study is to examine the influence of a brief post-session battery, designed to foster patient self-monitoring and reflection on their emotional reactions toward their psychotherapist, on the quality of the therapeutic relationship and treatment outcomes. Using an observational randomized control trial design, participants will be allocated into intervention and control groups. Those in the intervention group will complete a postsession battery following each therapy session, while the control group will only undergo regular treatment. Data collection will be facilitated through the Qualtrics online survey software and span baseline, mid-trial (5th week), and end-of-trial (10th week) assessments.

ELIGIBILITY:
Inclusion Criteria:

* being aged 18 years or older,
* being fluent in English,
* being currently under individual psychotherapy with a minimum frequency of two sessions per month.

Exclusion Criteria:

* having a legal guardian.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Outcomes in Routine Evaluation-Outcome Measure (Total score) from baseline to 5 weeks | Baseline, 5 weeks
  Measure of psychological distress devised to be administered during a course of psychotherapeutic treatment to determine treatment response. The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a 34-item self-report measure of change in psychotherapy. Total score ranges 0-136. Higher scores represent poorer overall functioning.
Change in Clinical Outcomes in Routine Evaluation-Outcome Measure (Total score) from baseline to 10 weeks | Baseline, 10 weeks
  Measure of psychological distress devised to be administered during a course of psychotherapeutic treatment to determine treatment response. The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a 34-item self-report measure of change in psychotherapy. Total score ranges 0-136. Higher scores represent poorer overall functioning.
Change in Clinical Outcomes in Routine Evaluation-Outcome Measure (Total score) from 5 weeks to 10 weeks | 5 weeks, 10 weeks.
  Measure of psychological distress devised to be administered during a course of psychotherapeutic treatment to determine treatment response. The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a 34-item self-report measure of change in psychotherapy. Total score ranges 0-136. Higher scores represent poorer overall functioning.
Change in Clinical Outcomes in Routine Evaluation-Outcome Measure (Subjective well-being deficits) from baseline to 5 weeks | Baseline, 5 weeks.
  Measure of psychological distress devised to be administered during a course of psychotherapeutic treatment to determine treatment response. The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a self-report measure of change in psychotherapy. The subjective well-being subscale score ranges 0-16). Higher scores represent poorer subjective well-being.
Change in Clinical Outcomes in Routine Evaluation-Outcome Measure (Subjective well-being deficits) from baseline to 10 weeks | Baseline, 10 weeks.
  Measure of psychological distress devised to be administered during a course of psychotherapeutic treatment to determine treatment response. The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a self-report measure of change in psychotherapy. The subjective well-being subscale score ranges 0-16). Higher scores represent poorer subjective well-being.
Change in Clinical Outcomes in Routine Evaluation-Outcome Measure (Subjective well-being deficits) from 5 weeks to 10 weeks | 5 weeks, 10 weeks.
  Measure of psychological distress devised to be administered during a course of psychotherapeutic treatment to determine treatment response. The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a self-report measure of change in psychotherapy. The subjective well-being subscale score ranges 0-16). Higher scores represent poorer subjective well-being.
Change in Clinical Outcomes in Routine Evaluation-Outcome Measure (Problems/symptoms) from baseline to 5 weeks | Baseline, 5 weeks.
  Measure of psychological distress devised to be administered during a course of psychotherapeutic treatment to determine treatment response. The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a self-report measure of change in psychotherapy. The problems/symptoms subscale score ranges 0-48). Higher scores represent greater problems/symptoms.
Change in Clinical Outcomes in Routine Evaluation-Outcome Measure (Problems/symptoms) from baseline to 10 weeks | Baseline, 10 weeks.
  Measure of psychological distress devised to be administered during a course of psychotherapeutic treatment to determine treatment response. The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a self-report measure of change in psychotherapy. The problems/symptoms subscale score ranges 0-48). Higher scores represent greater problems/symptoms.
Change in Clinical Outcomes in Routine Evaluation-Outcome Measure (Problems/symptoms) from 5 weeks to 10 weeks | 5 weeks, 10 weeks.
  Measure of psychological distress devised to be administered during a course of psychotherapeutic treatment to determine treatment response. The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a self-report measure of change in psychotherapy. The problems/symptoms subscale score ranges 0-48). Higher scores represent greater problems/symptoms.
Change in Clinical Outcomes in Routine Evaluation-Outcome Measure (Life functioning difficulties) from baseline to 5 weeks | Baseline, 5 weeks.
  Measure of psychological distress devised to be administered during a course of psychotherapeutic treatment to determine treatment response. The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a self-report measure of change in psychotherapy. The life functioning difficulties subscale score ranges 0-48). Higher scores represent greater life functioning difficulties.
Change in Clinical Outcomes in Routine Evaluation-Outcome Measure (Life functioning difficulties) from baseline to 10 weeks | Baseline, 10 weeks.
  Measure of psychological distress devised to be administered during a course of psychotherapeutic treatment to determine treatment response. The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a self-report measure of change in psychotherapy. The life functioning difficulties subscale score ranges 0-48). Higher scores represent greater life functioning difficulties.
Change in Clinical Outcomes in Routine Evaluation-Outcome Measure (Life functioning difficulties) from 5 weeks to 10 weeks | 5 weeks, 10 weeks.
  Measure of psychological distress devised to be administered during a course of psychotherapeutic treatment to determine treatment response. The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a self-report measure of change in psychotherapy. The life functioning difficulties subscale score ranges 0-48). Higher scores represent greater life functioning difficulties.
Change in Clinical Outcomes in Routine Evaluation-Outcome Measure (Risk/harm) from baseline to 5 weeks | Baseline, 5 weeks.
  Measure of psychological distress devised to be administered during a course of psychotherapeutic treatment to determine treatment response. The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a self-report measure of change in psychotherapy. The risk/harm subscale score ranges 0-26). Higher scores represent greater risk/harm.
Change in Clinical Outcomes in Routine Evaluation-Outcome Measure (Risk/harm) from baseline to 10 weeks | Baseline, 10 weeks.
  Measure of psychological distress devised to be administered during a course of psychotherapeutic treatment to determine treatment response. The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a self-report measure of change in psychotherapy. The risk/harm subscale score ranges 0-26). Higher scores represent greater risk/harm.
Change in Clinical Outcomes in Routine Evaluation-Outcome Measure (Risk/harm) from 5 weeks to 10 weeks | 5 weeks, 10 weeks.
  Measure of psychological distress devised to be administered during a course of psychotherapeutic treatment to determine treatment response. The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a self-report measure of change in psychotherapy. The risk/harm subscale score ranges 0-26). Higher scores represent greater risk/harm.

SECONDARY OUTCOMES:
Real Relationship Inventory-Client-Short form (Total score) | Up to 10 weeks.
  Measure of the real relationship between a therapist and participant from the participant's viewpoint. The Real Relationship Inventory-Client-Short form (RRI-C-SF) is an 8-item self-report measure of the quality of the real relationship and includes two subscales: Genuineness and Realism, both of which represent closely related dimensions of authenticity and perceptual accuracy within the therapeutic relationship. Total score ranges 0-40. Higher scores represent better quality of the real relationship. It will be assessed at baseline, mid-trial (5 weeks), and end-of-trial (10 weeks).
Real Relationship Inventory-Client-Short form (Genuineness) | Up to 10 weeks.
  Measure of the real relationship between a therapist and participant from the participant's viewpoint. The Real Relationship Inventory-Client-Short form (RRI-C-SF) is an 8-item self-report measure of the quality of the real relationship and includes two subscales: Genuineness and Realism, both of which represent closely related dimensions of authenticity and perceptual accuracy within the therapeutic relationship. The Genuineness subscale (3 items) score ranges 0-20. Higher scores represent higher perceived genuineness. It will be assessed at baseline, mid-trial (5 weeks), and end-of-trial (10 weeks).
Real Relationship Inventory-Client-Short form (Realism) | Up to 10 weeks.
  Measure of the real relationship between a therapist and participant from the participant's viewpoint. The Real Relationship Inventory-Client-Short form (RRI-C-SF) is an 8-item self-report measure of the quality of the real relationship and includes two subscales: Genuineness and Realism, both of which represent closely related dimensions of authenticity and perceptual accuracy within the therapeutic relationship. The Realism subscale (4 items) score range 0-20. Higher scores represent higher perceived realism. It will be assessed at baseline, mid-trial (5 weeks), and end-of-trial (10 weeks).
Working Alliance Inventory-Short Revised (Total score) | Up to 10 weeks.
  Measure of the working alliance between a therapist and participant from the participant's viewpoint. The Working Alliance Inventory-Short Revised (WAI-SR) is a 12-item self-report measure of the quality of the working alliance and includes three subscales: goal, task, and bond. Total score ranges 0-72. Higher scores indicate a stronger alliance. It will be assessed at baseline, mid-trial (5 weeks), and end-of-trial (10 weeks).
Working Alliance Inventory-Short Revised (Goal) | Up to 10 weeks.
  Measure of the working alliance between a therapist and participant from the participant's viewpoint. The Working Alliance Inventory-Short Revised (WAI-SR) is a 12-item self-report measure of the quality of the working alliance. The Goal subscale (3 items) score ranges 0-18. Higher scores indicate a stronger agreement on the tasks of therapy. It will be assessed at baseline, mid-trial (5 weeks), and end-of-trial (10 weeks).
Working Alliance Inventory-Short Revised (Task) | Up to 10 weeks.
  Measure of the working alliance between a therapist and participant from the participant's viewpoint. The Working Alliance Inventory-Short Revised (WAI-SR) is a 12-item self-report measure of the quality of the working alliance. The Task subscale score (3 items) ranges 0-18. Higher scores indicate a stronger agreement on the tasks of therapy. It will be assessed at baseline, mid-trial (5 weeks), and end-of-trial (10 weeks).
Working Alliance Inventory-Short Revised (Bond) | Up to 10 weeks.
  Measure of the working alliance between a therapist and participant from the participant's viewpoint. The Working Alliance Inventory-Short Revised (WAI-SR) is a 12-item self-report measure of the quality of the working alliance. The Bond subscale score (3 items) ranges 0-18. Higher scores indicate a stronger affective bond between the patient and the therapist. It will be assessed at baseline, mid-trial (5 weeks), and end-of-trial (10 weeks).
Number of sessions missed or canceled | Up to 10 weeks.
  Number of scheduled psychotherapy sessions that have been missed or canceled by the participant. It will be assessed at baseline, mid-trial (5 weeks), and end-of-trial (10 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Stefana, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Researchforme.Unc.Edu, Chapel Hill, North Carolina
  - Researchmatch.Org, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The Study protocol article will be published before data collection completion. Deidentified individual data that supports the results will be shared beginning 9 to 36 months following the publication of the research reports.
Access Criteria: Investigator has approved IRB, IEC), or REB and an executed data use/sharing agreement with the University of North Carolina at Chapel Hill.

REFERENCES:
- [Derived] Stefana A, Fusar-Poli P, Vieta E, Youngstrom EA. Effectiveness of a Novel Web-Based Intervention to Enhance Therapeutic Relationships and Treatment Outcomes in Adult Individual Psychotherapy: Randomized Controlled Trial and Analysis of Predictors of Dropouts. JMIR Ment Health. 2024 Nov 27;11:e63234. doi: 10.2196/63234. PMID 39602203
- [Derived] Stefana A, Vieta E, Fusar-Poli P, Youngstrom EA. Enhancing Psychotherapy Outcomes by Encouraging Patients to Regularly Self-Monitor, Reflect on, and Share Their Affective Responses Toward Their Therapist: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Apr 8;13:e55369. doi: 10.2196/55369. PMID 38587881